CLINICAL TRIAL: NCT05856409
Title: Clinical Application of 68Ga-FAPI PET Imaging in Detection of Ovarian Cancer Recurrence
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: LY2023-024-B
Record Dates: First submitted 2023-04-17; First posted 2023-05-12 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: 68Ga-FAPI; Ovarian Cancer; Epithelial Ovarian Cancer; Positron Emission Tomography
Keywords: 68Ga-FAPI; PET; ovarian cancer; recurrence detection
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Surgical or biopsy tumor tissue specimens
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: 68Ga-FAPI — [68Ga]-FAPI is tumor imaging agent for use with Positron Emission Tomography (PET) imaging for the detection of Fibroblast Activation Protein (FAP) positive cancer cells and cancer-associated fibroblasts (CAF)

SUMMARY:
This is a prospective study to investigate the potential efficacy of 68Ga-FAPI PET/CT for recurrence detection of epithelial ovarian cancer in comparison with 18F-FDG PET/CT.

DETAILED DESCRIPTION:
Gallium 68-labeled fibroblast-activation protein inhibitor (68Ga-FAPI) has recently been a potential radiotracer for gynecological malignancies,including ovarian cancer. Early detection and localization of sites of recurrence helps to identify ovarian cancer patients who will benefit the most from secondary surgery, chemotherapy, or radiation therapy. Its clinical utility for recurrence detection of epithelial ovarian cancer and histological validation of FAPI findings is not well established.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (age>18 and<80 years)
* patients with clinically suspected recurrent ovarian cancer
* patients who underwent paired 18F-FDG and 68Ga-FAPI PET/CT for the most proper treatment strategy within 1 week
* patients who did not receive any other treatment 4 weeks before PET imaging

Exclusion Criteria:

* pregnant patients
* patients with poor performance status
* patients unwilling to provide written informed consent

Ages: 18 Years to 80 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: A prospective cohort of patients with clinically suspected recurrent ovarian cancer were enrolled, who underwent paired 68Ga-FAPI and 18F-FDG PET/CT.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-05-10 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Performance | 1 year
  Sensitivity and Specificity of 68Ga-FAPI PET/CT for recurrence in comparison with 18F-FDG PET/CT
Maximum standardized uptake value（SUVmax） | 1 year
  Measurement of the maximum standardized uptake value of the lesion
Tumor-to-background ratio (TBR) | 1 year
  TBR was calculated according to the formula：TBR=SUVmax of lesion/SUVmax of background

SECONDARY OUTCOMES:
Correlation between FAPI expression and SUV in PET | 1 year
  Correlation between 68Ga-FAPI PET uptake intensity and histopathologic FAP expression. Validation via immunohistochemical FAP staining of pathological specimen

CONTACTS AND LOCATIONS:
Overall Officials: Jianjun Liu, PH.D, Principal Investigator — Ren Ji Hospital, School of Medicine, Shanghai Jiao Tong University
Locations (1):
- Ren Ji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No